CLINICAL TRIAL: NCT05199961
Title: Quality of Life of Adults With Diffuse Large B-cell Lymphoma Treated With Tisagenlecleucel
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor requested early termination
Sponsor: Pack Health (Industry)
Collaborators: Novartis (Industry); Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021C0141
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Quality of Life; Digital Health Coaching; adult; Receptors, Chimeric Antigen
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Intervention Model Description: A single cohort of up to 100 individuals receiving chimeric antigen receptor T cell therapy will be enrolled in the study, all of which will be enrolled in a 6-month digital health coaching program. Individuals will be enrolled at The Ohio State University Comprehensive Cancer Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Cohort Receiving Digital Health Coaching (Experimental): A single cohort of up to 100 individuals receiving chimeric antigen receptor T cell therapy will be enrolled in the study, all of whom will be enrolled in a 6-month digital health coaching program. Individuals will be enrolled at The Ohio State University Comprehensive Cancer Center.
  Interventions: Behavioral: Digital Health Coaching

INTERVENTIONS:
Behavioral: Digital Health Coaching — The digital health coaching program consists of weekly calls and delivery of evidence-based content across health and wellness domains (e.g. nutrition, exercise, physical, emotional and financial health) up to 4 times weekly via text, email or mobile application. The program is 6-months in duration and designed for engagement following CAR T cell infusion.

SUMMARY:
The aim of this non-interventional multi-center study is to evaluate quality of life (QOL) and other patient reported outcomes (PROs) among adults with diffuse large b-cell lymphoma (DLBCL) following Chimeric Antigen Receptor (CAR) T-cell therapy with tisagenlecleucel (Kymriah). Up to 100 individuals will be enrolled prior to tisagenlecleucel infusion in either the inpatient or ambulatory setting and followed for 6 months post-enrollment to evaluate changes in QOL from baseline to post-treatment, as measured by the Functional Assessment of Cancer Treatment- lymphoma (FACT-Lym). Secondary outcomes will assess patient self-efficacy in assessing for and managing treatment-related toxicities including cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) and communicating these and other concerns across care settings. To support patients and facilitate the collection of key PROs, a digital health coaching solution provided by Pack Health will be provided to each participant over the 6-month study enrollment. The digital coaching program provides an evidence-based curriculum focused on monitoring and managing CAR T-cell associated toxicities, enhancing overall wellness post-treatment, and navigating within and between referring and treating facilities. The participating site(s) will collect longitudinal PRO data focused on QOL across physiologic and psychosocial domains that coaching personnel will access and review with participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Able to read, speak and consent in English
* Diagnosis of diffuse large b-cell lymphoma
* Confirmed treatment with tisagenlecleucel (Kymriah)
* Internet access via smartphone, tablet, a computer, or another device with the capacity to receive calls, texts, or e-mails, as well as the electronic study assessments.

Exclusion Criteria:

* Individuals who are terminally ill, defined as individuals identified by their physician as likely having 6 months or less to live, or those individuals transitioned to comfort measures only (meaning only supportive care measures without curative focused treatment)
* Individuals for whom there is documentation of inability to provide consent in the medical record

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy- Lymphoma (FACT-Lym) | Change across Enrollment, Months 1,2,3,4,5,6
  The FACT-lym is a 42-item assessment that measures self-reported quality of life across 4 domains: physical, functional, emotional and social and includes 15 additional items validated specifically for individuals with lymphoma. The instrument can be scored as a whole as well as within the individual domains.

SECONDARY OUTCOMES:
SF-36 | Enrollment, Months 3,6
  The SF-36 is a validated measure for the assessment of health-related quality of life for individuals with diverse chronic conditions, including individuals with hematologic malignancies. It consists of 36-items assessing 8 health domains, including physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health. The instrument is scored on a scale of 0-100 for each of the 8 health domains. It was recently used in a study of quality-of-life following treatment with tisagenlecleucel.
Cancer Behavior Inventory- Brief (CBI-B) | Enrollment, Months 1,2,3,4,5,6
  This 12-item instrument measures self-efficacy in coping with cancer across 7 domains. These include: Seeking and Understanding Medical Information, Emotion Regulation, Coping with Treatment Related Side Effects, Accepting Cancer/ Maintaining a Positive Attitude, Seeking Social Support, and Using Spiritual Coping. The instrument utilizes a 9-point response scale ranging from 1 "Not at all confident" to 9 "Confident".
Subjective Assessment of Patient Experience in Managing CAR T Specific Care | Enrollment, Months 1,2,3,4,5,6
  As there are no currently validated instruments specific to CAR T-cell therapy, a 5-item assessment of patients' experience in monitoring, managing, and reporting treatment related toxicities will be created specifically for use in this study and will mirror the response scale in the CBI-B. This includes a 9-point response scale ranging from 1 "Not at all confident" to 9 "Confident". The following items will be included: 1) Understand the treatment toxicities I may experience while receiving CAR T-cell therapy; 2) Identify the signs and symptoms of these toxicities; 3) Communicate symptoms to provider; 4) Manage symptoms according to provider's instructions; 5) Explain treatment to a healthcare provider

OTHER OUTCOMES:
Socio-demographic, clinical, and treatment characteristics | Through study completion, at month 6
  Age, Race, Ethnicity, Sex at Birth, Gender Identity, Diagnosis, Treatment History, Co-morbid conditions, referring provider/institution, provider/institution for follow-up care, setting of CAR T-cell infusion
Digital Engagement | Through study completion, at month 6
  Frequency, types and duration of engagement with the digital health coaching platform
Treatment Response | Months 3,6
  Complete response, partial response, stable disease, progressive disease, unknown/not evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen McNally, PhD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buitrago J, Adkins S, Hawkins M, Iyamu K, Oort T. Adult Survivorship: Considerations Following CAR T-Cell Therapy. Clin J Oncol Nurs. 2019 Apr 1;23(2):42-48. doi: 10.1188/19.CJON.S1.42-48. PMID 30880816
- [Background] Chakraborty R, Sidana S, Shah GL, Scordo M, Hamilton BK, Majhail NS. Patient-Reported Outcomes with Chimeric Antigen Receptor T Cell Therapy: Challenges and Opportunities. Biol Blood Marrow Transplant. 2019 May;25(5):e155-e162. doi: 10.1016/j.bbmt.2018.11.025. Epub 2018 Nov 28. PMID 30500439
- [Background] Beaupierre A, Lundberg R, Marrero L, Jain M, Wang T, Alencar MC. Management Across Settings: An Ambulatory and Community Perspective for Patients Undergoing CAR T-Cell Therapy in Multiple Care Settings. Clin J Oncol Nurs. 2019 Apr 1;23(2):27-34. doi: 10.1188/19.CJON.S1.27-34. PMID 30880815
- [Background] Ventura F, Ohlen J, Koinberg I. An integrative review of supportive e-health programs in cancer care. Eur J Oncol Nurs. 2013 Aug;17(4):498-507. doi: 10.1016/j.ejon.2012.10.007. Epub 2012 Nov 15. PMID 23158437
- [Background] Madore S, Kilbourn K, Valverde P, Borrayo E, Raich P. Feasibility of a psychosocial and patient navigation intervention to improve access to treatment among underserved breast cancer patients. Support Care Cancer. 2014 Aug;22(8):2085-93. doi: 10.1007/s00520-014-2176-5. Epub 2014 Mar 18. PMID 24639035
- [Background] Jansen F, van Uden-Kraan CF, van Zwieten V, Witte BI, Verdonck-de Leeuw IM. Cancer survivors' perceived need for supportive care and their attitude towards self-management and eHealth. Support Care Cancer. 2015 Jun;23(6):1679-88. doi: 10.1007/s00520-014-2514-7. Epub 2014 Nov 26. PMID 25424520
- [Background] Green AC, Hayman LL, Cooley ME. Multiple health behavior change in adults with or at risk for cancer: a systematic review. Am J Health Behav. 2015 May;39(3):380-94. doi: 10.5993/AJHB.39.3.11. PMID 25741683
- [Background] Girault A, Ferrua M, Lalloue B, Sicotte C, Fourcade A, Yatim F, Hebert G, Di Palma M, Minvielle E. Internet-based technologies to improve cancer care coordination: current use and attitudes among cancer patients. Eur J Cancer. 2015 Mar;51(4):551-557. doi: 10.1016/j.ejca.2014.12.001. Epub 2015 Feb 4. PMID 25661828
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Maziarz RT, Waller EK, Jaeger U, Fleury I, McGuirk J, Holte H, Jaglowski S, Schuster SJ, Bishop MR, Westin JR, Mielke S, Teshima T, Bachanova V, Foley SR, Borchmann P, Salles GA, Zhang J, Tiwari R, Pacaud LB, Ma Q, Tam CS. Patient-reported long-term quality of life after tisagenlecleucel in relapsed/refractory diffuse large B-cell lymphoma. Blood Adv. 2020 Feb 25;4(4):629-637. doi: 10.1182/bloodadvances.2019001026. PMID 32074277
- [Background] Bunevicius A. Reliability and validity of the SF-36 Health Survey Questionnaire in patients with brain tumors: a cross-sectional study. Health Qual Life Outcomes. 2017 May 4;15(1):92. doi: 10.1186/s12955-017-0665-1. PMID 28472964
- [Background] Hlubocky FJ, Webster K, Beaumont J, Cashy J, Paul D, Abernethy A, Syrjala KL, Von Roenn J, Cella D. A preliminary study of a health related quality of life assessment of priority symptoms in advanced lymphoma: the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy - Lymphoma Symptom Index. Leuk Lymphoma. 2013 Sep;54(9):1942-6. doi: 10.3109/10428194.2012.762977. Epub 2013 Feb 7. PMID 23320888
- [Background] Heitzmann CA, Merluzzi TV, Jean-Pierre P, Roscoe JA, Kirsh KL, Passik SD. Assessing self-efficacy for coping with cancer: development and psychometric analysis of the brief version of the Cancer Behavior Inventory (CBI-B). Psychooncology. 2011 Mar;20(3):302-12. doi: 10.1002/pon.1735. PMID 20878830
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- See also: FDA approves tisagenlecleucel for adults with relapsed or refractory large B-cell lymphoma — https://www.fda.gov/drugs/resources-information-approved-drugs/fda-approves-tisagenlecleucel-adults-relapsed-or-refractory-large-b-cell-lymphoma